CLINICAL TRIAL: NCT05202301
Title: Medication Adherence and Discontinuation Among Patients With Prostate Cancer Who Initiated Second Generation Androgen Receptor Inhibitors
Brief Title: A Study Using Available Data to Learn to What Extent Patients With Prostate Cancer Who Received Second Generation Androgen Receptor Inhibitors Took Their Medication as Prescribed or Stopped Taking Their Medication Completely
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 22053
Record Dates: First submitted 2022-01-10; First posted 2022-01-21 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — darolutamide; enzalutamide; apalutamide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Darolutamide cohort (Daro): Participants received Second Generation Androgen Receptor Inhibitor (SGARI) Darolutamide as initial treatment
  Interventions: Drug: Darolutamide (Nubeqa, BAY1841788)
- Enzalutamide cohort (Enza): Participants received Second Generation Androgen Receptor Inhibitor (SGARI) Enzalutamide as initial treatment
  Interventions: Drug: Enzalutamide
- Apalutamide cohort (Apa): Participants received Second Generation Androgen Receptor Inhibitor (SGARI) Apalutamide as initial treatment
  Interventions: Drug: Apalutamide

INTERVENTIONS:
Drug: Darolutamide (Nubeqa, BAY1841788) — Retrospective cohort analysis, using the IQVIA Real-World Data Adjudicated Claims, US claims database
  Groups: Darolutamide cohort (Daro)
Drug: Enzalutamide — Retrospective cohort analysis, using the IQVIA Real-World Data Adjudicated Claims, US claims database
  Groups: Enzalutamide cohort (Enza)
Drug: Apalutamide — Retrospective cohort analysis, using the IQVIA Real-World Data Adjudicated Claims, US claims database
  Groups: Apalutamide cohort (Apa)

SUMMARY:
This is an observational study in which patient data from the past on men with prostate cancer are studied.

Cancer is a condition in which the body cannot control the growth of cells and tumors may form. If tumors form in the prostate, male sex hormones (androgens) can sometimes help the cancer spread and grow. Cancer that spreads to other parts of the body is called metastasis.

Androgens are mainly made in the testicles. There are treatments available for men with prostate cancer to lower the levels of these hormones in the body. These treatments are called androgen deprivation therapy (ADT). Some men with prostate cancer respond to ADT, but in some cases, prostate cancer may overcome the therapy and worsen despite low androgens levels.

Second generation androgen receptor inhibitors (SGARIs) including darolutamide, apalutamide, and enzalutamide are available for the treatment of prostate cancer in addition to ADT. SGARIs work by blocking androgens from attaching to proteins in cancer cells in the prostate.

Clinical studies have shown that men with prostate cancer benefit from these treatments. But besides benefits, unfavorable reactions related to these treatments also influence which treatment is chosen, if the treatment is taken as intended or if it is even stopped.

Unfavorable reactions observed for darolutamide, apalutamide, and enzalutamide differ from each other. In clinical trials, severe unfavorable reactions occurred less often for darolutamide.

But information on how unfavorable reactions of each treatment influence their intake in actual or "real-world" prostate cancer treatment is missing.

The main aim of this observational study is to learn to what extent SGARI treatments are taken as prescribed and how often their intake is completely stopped. To find this out, researchers will collect available treatment data of adult men with prostate cancer from the United States who started SGARI treatments between August 2019 and March 2021. The data will be drawn from the IQVIA database.

For each man, data from up to 1 year prior SGARI treatment until at least 3 months after treatment start (up to the 30 June 2021) will be collected.

The researchers will look at the percentage of men who:

* completely stopped to take their treatment or
* took the treatment as prescribed.

The results for each treatment (darolutamide, apalutamide, and enzalutamide) will then be compared to find possible differences.

There will be no required visits with a study doctor or required tests in this study since only patient data from the past are studied.

ELIGIBILITY:
Inclusion Criteria:

* Have at least 1 prescription claims for enzalutamide (National Drug Code [NDC]: 00469-0125-99, 00469-0625-99, 00469-0725-60), apalutamide (NDC: 59676-600-12, 59676-600-56, 59676-600-99) or darolutamide (NDC: 50419-395-01, 50419-395-72) during the index identification period.

  -- The date of the earliest SGARI claim to occur during this period will be defined as the index date with the corresponding SGARI as the index treatment.
* Have ≥1 diagnosis of prostate cancer (ICD-10 code C61.) during the overall baseline period.
* Age ≥18 years and male gender on the index date.
* Have continuous health plan enrollment with medical and pharmacy benefits for at least 6 months prior to the index date.
* Have continuous health plan enrollment with medical and pharmacy benefits for at least 3 months after the index date and throughout the follow-up period.

Exclusion Criteria:

* Since patients should not be prescribed more than one SGARI when initiating treatment, patients with more than one SGARI prescribed on the index date will be excluded from the study. This will allow each patient to be assigned to a single study cohort.
* In order to select patients who are initiating SGARI treatment, patients with the index SGARI treatment during the 1 year baseline period will be excluded from the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed with Prostate Cancer who newly initiate Second Generation Androgen Receptor Inhibitors treatment in United States from 01 Aug 2019 to 31 Mar 2021.
Sampling Method: Non-Probability Sample
Enrollment: 13779 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Discontinuation rate of SGARI treatment | Retrospective analysis from index date 01-Aug-2019 up to 30-Jun-2021
  The proportion of patients who discontinue their index SGARI treatment at 3 months, 6 months, 1 year and acutely (discontinuation within 90 days) will be evaluated. In addition, time to discontinuation will be assessed.
  Discontinuation will be defined as a gap of ≥60 days from the end of the days of supply (DOS) of a prescription claim for the index SGARI to the date of the next prescription claim. The date of the last day of supply for the prescription claim that occurs immediately prior to the gap will be defined as the date of discontinuation.
  Discontinuation rate will be defined as the proportion of patients with discontinuation within a set time period (3 months, 6 months, 1 year).
Time to discontinuation (days) of SGARI treatment | Retrospective analysis from index date 01-Aug-2019 up to 30-Jun-2021
  Time to discontinuation will be assessed over the entire observation period
Adherence of SGARI treatment | Retrospective analysis from index date 01-Aug-2019 up to 30-Jun-2021
  Medication adherence will be assessed using medication possession ratio (MPR) and proportion of days covered (PDC)

SECONDARY OUTCOMES:
Treatment duration of SGARI treatment | Retrospective analysis from index date 01-Aug-2019 up to 30-Jun-2021
  Continuous treatment duration will be defined as the number of days from the index date to the date of discontinuation or the censoring date, whichever is earlier
Risk factors for treatment discontinuation | Retrospective analysis from index date 01-Aug-2019 up to 30-Jun-2021
  Sociodemographic and clinical patient characteristics will be assessed to identify risk factors associated with the discontinuation of index SGARI treatment using multivariable logistic regression models.
The proportion of patients who had evidence of dose modification of their index SGARI treatment | Retrospective analysis from index date 01-Aug-2019 up to 30-Jun-2021
  Dose modifications will be measured using relative dose intensity (RDI) calculated as the ratio of the delivered dose intensity to the standard dose intensity as recommended for each SGARI
Time to first dose modification (days) of index SGARI treatment | Retrospective analysis from index date 01-Aug-2019 up to 30-Jun-2021
Descriptive summary of the baseline demographics of Prostate Cancer (PC) patients treated with SGARIs | Retrospective analysis during index identification period, from 01-Aug-2018 up to 31-Mar-2021
  Patient demographics evaluated on the index date will consist of age, race, region, insurance and health plan type when available
Descriptive summary of the Comorbid conditions | Retrospective analysis from 01-Aug-2018 up to 31-Mar-2021
  For each qualified patient, the twelve-month baseline period or on the index date will be examined in order to compile patient histories
Descriptive summary of the Charlson Comorbidity Index (CCI) | Retrospective analysis from 01-Aug-2018 up to 31-Mar-2021
  Charlson Comorbidity Index (CCI): The CCI is a method of estimating the one-year mortality for a patient with certain comorbid conditions. Each comorbid condition is given a score of 1, 2, 3 or 6 based on the degree of mortality attributed to the condition. The scores are summed to yield a total index score which can be used to predict long-term survival. The CCI will be calculated for each patient based on all diagnoses during the 1 year baseline period and the index date
The proportion of patients who received different PC related medications | Retrospective analysis from 01-Aug-2018 up to 30-Jun-2021
  PC related medications: Androgen Deprivation Therapy (ADT) alone; First-generation antiandrogens; Second-generation androgen receptor inhibitors (SGARI); Chemotherapy; Other chemotherapy; Immunotherapy; Bone health agents; Radiopharmaceutical
Descriptive summary of the baseline SGARI-class exposure status | Retrospective analysis from 01-Aug-2018 up to 31-Mar-2021
  SGARI-class exposure status: SGARI-class naïve; SGARI-class experienced
Descriptive summary of the baseline Hormone sensitivity status | Retrospective analysis from 01-Aug-2018 up to 31-Mar-2021
  Hormone sensitivity status: Hormone-sensitive PC; Castration-resistant PC; Unknown

CONTACTS AND LOCATIONS:
Locations (1):
- Bayer, Whippany, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.